CLINICAL TRIAL: NCT04886440
Title: Predictive Value of the Sialendoscopy in Treatment of Submandibular Gland Sialolithiasis: a Retrospective Study
Brief Title: Sialendoscopy in Treatment of Submandibular Gland Sialolithiasis
Acronym: SIAGLA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01Obs-CHRMT
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Lithiasis
Keywords: sialendoscopy; submandibular gland; classification
MeSH Terms: conditions — Lithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Salivary disorders are common reason for ENT specialist consultation. Sialolithiasis are the most frequent salivary obstruction disease and are characterized by the development of calcified structures in the salivary gland, especially in the submandibular gland.

The management of salivary obstruction has changed over the past 30 years. Sialendoscopy is considered as a minimally invasive procedure that allows endoscopic visualization of the salivary ductal system and is increasingly used in both diagnosis and treatment. Moreover, many studies have shown the effectiveness of this procedure.

Classification of lithiasis has been set up in 2008 to standardize the nomenclature and was used for patient care since 2009. The main objective of this study is to evaluate the relevance of the lithiasis's classification to predict the efficacy of sialendoscopy in treatment of sialolithiases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient treated in CHR Metz-Thionville between 2013 and 2020
* With a pathological impairment (suspected or confirmed) of a salivary gland
* With sialendoscopy indication for diagnosis and/or treatment

Exclusion Criteria:

* Opposed to use data
* Without sialendoscopy indication
* Without lithiasis salivary gland disorder
* With parotid gland lithiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with submandibular sialolithiasis
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Recurrence of symptom | Month 6
  Absence or presence of symptoms associated to lithiasis

SECONDARY OUTCOMES:
Number of clinical signs | Day 1
  number of clinical signs of the clinical suspicion
Number of intraoperative complications | Day 1
  number of intraoperative complications
Number of post-operative complications | Day 1
  Number of post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France